CLINICAL TRIAL: NCT02295046
Title: Open Label, Randomized, Two-treatment, Two-period, Two-sequence,Crossover, Single Dose, Oral Bioequivalence Study of Amlodipine Besylate/Atorvastatin Calcium Tablets 10mg/80mg Under Fasting Condition
Brief Title: Bioavailability Study of Amlodipine Besylate/Atorvastatin Calcium Tablets 10/80 mg Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AMAT-BESD-03-RDL/10
Record Dates: First submitted 2014-11-17; First posted 2014-11-19 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2011-12

CONDITIONS: Healthy
MeSH Terms: interventions — Amlodipine; Atorvastatin; amlodipine, atorvastatin drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amlodipine besylate/Atorvastatin calcium tablets 10/80 mg (Experimental): Amlodipine besylate/Atorvastatin calcium tablets 10/80 mg of Dr. Reddys Laboratories Limited
  Interventions: Drug: Amlodipine besylate/Atorvastatin calcium
- Caduet (Active Comparator): Caduet® 10/80 mg tablets of Pfizer, Ireland
  Interventions: Drug: Amlodipine besylate/Atorvastatin calcium

INTERVENTIONS:
Drug: Amlodipine besylate/Atorvastatin calcium — Amlodipine besylate/Atorvastatin calcium 10/80 mg
  Other Names: Caduet

SUMMARY:
This study is to assess the bioequivalence between Amlodipine besylate/Atorvastatin calcium Tablets 10mg/80mg of Dr. Reddy's Laboratories Limited, India and CADUET® (amlodipine besylate and atorvastatin calcium) tablets 10mg/80mg of Pfizer Ireland Pharmaceuticals Dublin, Ireland in Healthy Male and Female Volunteers under Fasting conditions.

DETAILED DESCRIPTION:
Open label, randomized, two-treatment, two-period, two-sequence, crossover, single dose, oral bioequivalence study of Amlodipine besylate/Atorvastatin calcium Tablets 10mg/80mg under Fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female volunteers between 18 and 55 years of age
2. Subject with the Body Mass Index within 18.5 and 24.9 kg/m2, weight not less than 50 kg
3. Normal health as determined by personal medical history, haematology, clinical chemistry and urinalysis laboratory profiles
4. Non smokers or ex-smokers that gave up smoking for at least two years prior to the study
5. The subject agrees to abstain from alcohol, food and drinks containing methylxanthines (tea, cola, chocolate) for 48 hours prior to study drug administration and during each study period and from grapefruit-containing food and beverages for 48 hours prior to study drug administration and during each study period
6. Ability to understand the full nature and purpose of the study, including possible risks and side effects; ability to cooperate with the Clinical Investigator and to comply with the requirements of the entire study
7. Informed written consent given voluntary before the initiation of the pre-study screening
8. Negative results to the HIV, hepatitis C or hepatitis B test
9. Negative results from pregnancy tests (for female subjects only)
10. Non-lactating woman (for female subjects only)
11. Subjects using non-hormonal contraceptive measures during the study (for female subjects only)
12. Normal creatine phosphokinase (CPK) levels at the time of check-in of each period.

Exclusion Criteria:

1. History of hypersensitivity to the test drug (Amlodipine Besylate/Atorvastatin Calcium) or to drugs belonging to the same pharmacological and chemical class and inactive ingredients of the formulation
2. Participation in a clinical study with an investigational product in the preceding three months or in a clinical study with a generic product in the preceding two months
3. Hospitalization for any reason within eight weeks prior to the study initiation
4. Donation of 450 ml or more of blood, within eight weeks prior to the study initiation
5. Intake of any prescription or non-prescription drug (including anti-acids, analgesics, statins, cyclosporin, fibric acid derivatives, erythromycin, azole antifungals, niacin, oral contraceptives etc.) during the two weeks preceding the study or throughout the study
6. History of presence of any relevant medical condition including cancer, significant disease of the renal, hepatic, immunological, dermatological, gastrointestinal, respiratory, cardiovascular, endocrine or locomotor systems, and any metabolic, haematological neurological disorder or psychiatric disorder
7. History or presence of drug or alcohol abuse, within the past year
8. History or any current condition or other disease known to interfere with the absorption, distribution, metabolism or excretion of investigational medicines
9. ECG having evidence of clinically significant abnormalities
10. Presence of any acute or chronic infectious disease
11. Positive results to the HIV, hepatitis C or hepatitis B tests
12. Positive results to the breath alcohol test and drugs of abuse checks
13. Positive results to the pregnancy tests (for female subjects only)
14. Subject is vegetarian or follows particular diets
15. A history of difficulty with donating blood.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2011-10; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Area under curve (AUC) | 0.50; 1.00; 2.00; 3.00; 4.00; 5.00; 6.00; 7.00; 8.00; 10.00; 11.00; 12.00 16.00; 24.00; 36.00;48.00 and 72.00 hours post dose for Amlodipine

SECONDARY OUTCOMES:
Area under curve (AUC) | 10 min; 20 min; 30 min; 40 min; 50 min; 1.00; 1.25; 1.50; 1.75; 2.00; 2.25; 2.50; 2.75; 3.00; 3.50; 4.00; 4.50; 5.00; 6.00; 8.00; 10.00; 12.00 16.00;24.00; 36.00; 48.00 and 72.00 hours post dose for Atorvastatin

CONTACTS AND LOCATIONS:
Overall Officials: Dr. V Parasca, MD, Principal Investigator — 3S-Pharmacological Consultation & Research GmbH
Locations (1):
- 3S-Pharmacological Consultation & Research GmbH, D-27243 Harpstedt, Koenigsberger, Germany